CLINICAL TRIAL: NCT06805799
Title: Maternal-Infant Stress Reactivity as an Intergenerational Pathway to Cardiovascular Disease Risk
Brief Title: Stress Reactivity and Mother-Infant Cardiovascular Disease Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Micheline Anderson, Assistant Professor of Psychiatry and Human Behavior, Lifespan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1679889-63; 5U54GM115677-09 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-02-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Maternal Health; Infant Health; Hypertension; Behavioral Medicine; Mindfulness; Psychophysiology; Cardiovascular Diseases; Cardiovascular Diseases Risk
Keywords: Mindfulness; Psychophysiology; Coregulation; Maternal-infant Coregulation; Cardiovascular Disease Risk; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a follow-up study to an RCT of prenatal mindfulness vs. TAU for pregnant women at risk for hypertensive disorder of pregnancy. At 6 months postpartum, all participants who consent to this follow-up study will engage with the Still Face Paradigm, a well-validated lab-based protocol that elicits behavioral and physiological reactivity from mother and infant. Individual and dyadic physiological reactivity will be examined in relation to mother and infant biomarkers of cardiovascular risk at 12 months postpartum. Self and dyadic participant responses to the SFP will then be compared by treatment arm (MT vs. TAU).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Follow-up to Mindfulness RCT Using Still Face Paradigm (Experimental): Postpartum people who participated in either a mindfulness arm or TAU during an RCT examining prenatal mindfulness for pregnant people at risk for hypertensive disorders of pregnancy and their infants at 6 months of age will attend one session in which they are consented and prepared for the Still Face Paradigm (application of electrodes and RSA monitors, placement of video equipment). The SFP consists of a sequence of three, 2-minute episodes in which the parent and the infant are seated about one meter away from each other. During the first episode, the parent is free to play with the infant as they would at home. During the "still-face" episode (SF), the parent maintains a neutral face and is told not to touch or interact with the infant. The third episode is a resumption of play sometimes referred to as the "reunion" episode.
  Interventions: Other: Follow up to Mindfulness RCT using a Still Face Paradigm

INTERVENTIONS:
Other: Follow up to Mindfulness RCT using a Still Face Paradigm — Mothers who participated in an RCT of mindfulness to prevent hypertensive disorders of pregnancy and their infants at 6 months of age will attend one session in which they are consented and prepared for the Still Face Paradigm (SFP). The SFP consists of a sequence of three, 2-minute episodes in which the parent and the infant are seated about one meter away from each other. Across a pre-task baseline, task episodes (free play and still-face), and recovery periods, mothers and infants will wear wireless heart rate monitors to assess respiratory sinus arrhythmia and heart rate. At 12 months, mothers will complete lab work to assess cardiovascular risk and infants' growth velocity will be culled from pediatric medical records.

SUMMARY:
Prenatal Mindfulness training (MT) shows promise as a preventive intervention against hypertensive disorders of pregnancy (HDP) and may reduce risk for offspring cardiovascular disease (CVD). One proposed mechanism of MT to reduced CVD risk is improved self-regulation following stress. Perhaps the most crucial contributor to the development of self-regulation in the first year is the psychophysiological coregulatory relationship between mother and infant. However, this self-and co-regulation among women exposed to prenatal MT has not been studied and has yet to be examined in relation to CVD risk. The goal of this proposed project is to evaluate maternal-infant physiological reactivity to and recovery from stress at 6 months postpartum following prenatal MT, and to examine the relationship between these maternal infant stress responses and maternal-infant CVD risk at 12 months postpartum.

Using a lab-based stress paradigm and well-validated biomarkers of mother and infant CVD risk, the investigators will assess respiratory sinus arrhythmia and heart rate at 6 months postpartum for 40 mother-infant dyads who have completed either prenatal MT or a usual care arm of an RCT examining MT for women at risk for HDP. The investigators will compare maternal, infant, and dyadic stress responses by treatment arm. Then, cardiac stress responses will be examined as predictors of maternal and infant biomarkers of CVD risk at 12 months postpartum.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP) affect 1 out of 10 pregnancies, contribute annually to over two billion dollars of health care utilization costs, and are a leading cause of maternal morbidity and mortality in the United States. HDP confer long-term cardiovascular disease (CVD) risk for both mother and infant. Thus, prevention of prenatal HDP is essential to reducing intergenerational transmission of CVD risk. Prenatal mindfulness training (MT) has shown promise as a non-pharmacological intervention to prevent HDP and is associated with improved mother-infant outcomes at birth. Benefits of prenatal MT on maternal-infant stress responses and concomitant effects on CVD risk have not been examined.

One proposed mechanism thought to confer cardiovascular benefits of MT is improved physiological stress response via the autonomic nervous system (ANS). ANS dysfunction has been linked with early childhood physical health concerns, such as obesity and elevated blood pressure, and increased CVD risk in adulthood, and thus may be a significant target for interventions aiming to disrupt intergenerational risk for CVD.There is emerging evidence that prenatal MT interventions may improve sympathetic reactivity to and recovery from stress (as measured by pre-ejection period activity) in 6-month old infants. Biobehavioral frameworks of attachment propose that mother-child dyads engage in physiological coregulation that influences self-regulatory processes. Maternal-infant synchrony of heartbeat and motor activity begins in utero and may promote children's physical and behavioral health. Concordance of maternal-infant self-regulation in stressful situations, a proxy of adaptive psychophysiological reactivity, may thus be associated with reduced CVD risk. However, it is not yet known whether prenatal MT is associated with improved maternal-infant regulation of ANS responses to stress, or whether these responses are associated with maternal and pediatric cardiovascular outcomes. These data are essential for the development of targeted parenting interventions that promote adaptive coregulatory stress responses and disrupt postpartum pathways for intergenerational CVD risk.

To address this knowledge gap, this study will examine effects of a prenatal MT intervention on postpartum maternal-infant psychophysiological coregulatory processes that may decrease maternal and infant CVD. The study will leverage the data and infrastructure from an ongoing RCT (PI: Mentor Bublitz; R01HL157288) examining mechanisms of a prenatal MT intervention on the prevention of HDP. At 6 months postpartum, maternal-infant physiological reactivity to stress will be assessed. At 12 months postpartum, maternal and infant CVD risk will be measured. This study aims to: 1) Evaluate psychophysiological responses to stress in women randomized to MT vs usual care and their offspring and 2) Evaluate the relationship between maternal-infant psychophysiological responses to stress and cardiovascular markers of disease risk. Using innovative assessment and analysis of self-and coregulation, results will provide insights into whether and how prenatal mindfulness impacts stress reactivity for mothers and their infants and, for the first time, whether coregulatory physiology is linked with cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* For the parent RCT study: Inclusion criteria: singleton pregnancy, English speaking, >18 years old, <20 weeks' gestation at enrollment, normotensive at enrollment, and criteria consistent with 'moderate' to 'high' risk for preeclampsia based on American College of Obstetrician and Gynecologist guidelines. For the current research study: Participants will be (n=40) individuals from the parent RCT who have consented to be contacted for future research in the parent study and are not pregnant during the mentored research study procedures.

Exclusion Criteria:

For the parent RCT study: Exclusion criteria: multiple gestations; chronic hypertension; active suicidality or psychosis; ongoing mind-body practice (e.g., yoga, meditation, mindfulness > once a week).

-

Min Age: 6 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maternal-Infant Stress reactivity | Single episode of assessment at 6 months postpartum
  Stress reactivity will be measured using respiratory sinus arrhythmia (RSA), collected during all phases of the Still Face Paradigm via wireless ECG monitors on both mothers and infants. Maternal-infant RSA synchrony value per 30-second epoch will be calculated using CardioBatch Plus Synchrony, which quantifies the amplitude of RSA with age-specific parameters that are sensitive to the maturational shifts in the frequency of spontaneous breathing, and is statistically equivalent to frequency domain methods (i.e., spectral analysis) for calculation of the amplitude of RSA when heart period data are stationary. RSA will be quantified during each sequential 30-s epoch within each condition of the SFP and then compared across treatment arms.

SECONDARY OUTCOMES:
Maternal cardiovascular risk biometrics | Single assessment at 12 months postpartum
  Biomarkers of Cardiovascular Risk. This study leverage CVD biomarkers from the parent RCT at 12 months postpartum to test associations with maternal-infant stress reactivity. Several CVD biomarkers in postpartum women will be assessed via maternal serum (total cholesterol, LDL, HDL, triglycerides, high sensitivity C-reactive protein, and insulin resistance (HOMA-IR) using standard laboratory procedures ambulatory blood pressure monitoring, and anthropometric data collection (BMI). Maternal CVD risk at 12 months postpartum will be quantified using a composite risk score (ranging from 0-8), consistent with the method chosen by the parent RCT and recommendations from the World Health Organization and other CVD risk calculators.
Infant cardiovascular risk biometrics | Single assessment at 12 months postpartum
  Birthweight, length, and gestational age at birth is being extracted from medical records during the parent study. Infant CVD Risk at 12 months of age will be measured by infant weight-for-length growth velocity (World Health Organization; z score) using these data.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Medicine Collaborative, Lifespan, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No